CLINICAL TRIAL: NCT02485470
Title: Benefits of MPACT in Locally Advanced Head and Neck Cancer Patients Undergoing Chemoradiotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2015.073; HUM00100889 (Other: University of Michigan)
Record Dates: First submitted 2015-06-26; First posted 2015-06-30 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MPACT (Experimental): A 7-week (7 weeks x 3 sessions per week), on site, functional resistance training (FRT) as well as a walking program concurrent with CCRT will be followed by a 7-week post-CCRT home program. The protocol follows American College of Sports Medicine (ACSM) prescription guidelines for cancer patients.
  Interventions: Other: MPACT
- Usual Care (No Intervention)

INTERVENTIONS:
Other: MPACT — Maintaining Physical Activity during Cancer Treatment
  Arms: MPACT

SUMMARY:
The goal of this study is to test, in a randomized controlled trial among head and neck cancer patients, the short and longer term effects of the MPACT (Maintaining Physical Activity during Cancer Treatment) program (infused with motivational interviewing and self-determination theory-based strategies) initiated at the time of concurrent chemotherapy with radiation (CCRT), on key outcomes such as functional mobility and quality of life, and ultimately physical activity. The central hypotheses is that in head and neck cancer patients undergoing CCRT, the MPACT program, as compared to usual care controls, will result in less acute decline, faster recovery, and better maintenance of these key outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than or equal to 40 years old with AJCC (American Joint Committee on Cancer) stage II-IV head and neck squamous cell carcinoma who are beginning first-line non-surgical treatment with concurrent chemoradiotherapy (CCRT) and who are capable of understanding and adhering to the protocol requirements
* Patients must be willing to comply with the study procedures and visits.

Exclusion Criteria:

* Active or symptomatic cardiopulmonary disease
* Substantial dementia
* Acute medical conditions, such as acute flare-up of joint condition or infection
* Participants must not be actively receiving physical therapy in a relevant area, at the time of enrollment, or participating in intensive (30 min per day) aerobic program three times per week.
* Patients are actively being treated for another cancer at the time of enrollment
* Active or unstable metabolic conditions such as brittle diabetes or severe anemia
* Alcohol intake less than 3 ounces per day
* Hemiplegia or lower limb amputation
* Significant orthopedic or musculoskeletal condition that does not allow weight bearing
* Unable to maintain safe stance and walk, either with or without an assistive device

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-02; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Mean change in 6 minute walk distance (6MWD) | 1 Year
  6 MWD will be assessed at baseline, at weeks 4, 7, 11, and 14 and at 6 months and 1 year. The change from baseline will be calculated for each participant and longitudinal mixed models will be used to characterize mean outcomes over time for each intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Mierzwa, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- The University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States